CLINICAL TRIAL: NCT04709640
Title: Tailored, Intervention to Improve Medication Management in Community-Dwelling Older Adults: A Pilot Study
Brief Title: Pilot Study to Improve Medication Management in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Susan Stark, Associate Professor of Occupational Therapy, Neurology and Social Work, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201708062
Record Dates: First submitted 2020-10-13; First posted 2021-01-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Medication Management Intervention (Experimental): This research study involved an initial 1.5 hour visit and 2-3 follow up home visits (each lasting 60 minutes). Participants received 2-3 home visits during which they received recommendations on strategies which will improve medication management. Level II occupational therapy fieldwork students made the recommendations, after approval from their supervising licensed OT. The OT fieldwork students provided assistance to the individual in implementing strategies, obtaining adaptive equipment at little or no cost to the individual.
  Interventions: Other: Tailored Medication Management Intervention

INTERVENTIONS:
Other: Tailored Medication Management Intervention — This research study involved an initial 1.5 hour visit and 2-3 follow up home visits (each lasting 60 minutes). Participants received 2-3 home visits during which they received recommendations on strategies which will improve medication management. Level II occupational therapy fieldwork students made the recommendations, after approval from their supervising licensed OT. The OT fieldwork students provided assistance to the individual in implementing strategies, obtaining adaptive equipment at little or no cost to the individual.

SUMMARY:
This pilot study seeks to determine the acceptability and feasibility of the intervention to improve ability of older adults to management medication with community dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* taking four or more prescription medications
* self-reported decreased medication adherence.

Exclusion Criteria:

* significant cognitive impairment as indicated by a score of 10 or more on the Short Blessed Test
* Resides in an institutionalized setting.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
In-Home Medication Management Evaluation (HOME-Rx) | 1 month
  The HOME-Rx is a performance-based tool designed to identify functional barriers to medication management for community-dwelling older adults. Its purpose is to identify common and specific barriers to independence in medication management for older adults living independently in the community. We will use the I-HOPE measure the severity of barriers impacting medication management before and after the intervention. We will also measure the performance and satisfication of the older adult to perform their medication management tasks independently before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No